CLINICAL TRIAL: NCT00202917
Title: Multicenter Phase I/II Study of Haploidentical Hematopoietic Cell Transplantation With CD3/CD19 Depleted Grafts in Patients With Treatment Refractory Hematologic Malignancies
Brief Title: Haploidentical Transplantation With CD3/CD19 Depleted Grafts in Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E203/2004; IRB Project Nr. 21/2004; HSZ-001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Hematologic Malignancies
Keywords: haploidentical transplantation; immunomagnetic cell sorting; allogeneic hematopoietic cell transplantation; dose reduced conditioning
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; Thiotepa; Melphalan

INTERVENTIONS:
Drug: Fludarabine
Drug: Thiotepa
Drug: Melphalan
Drug: OKT-3
Procedure: CD3/CD19 depletion on CliniMACS

SUMMARY:
The purpose of this study is to study the feasibility and Toxicity of allogeneic haploidentical hematopoietic cell transplantation with CD3/CD19 depleted stem cells and a dose reduced conditioning.

DETAILED DESCRIPTION:
Transplantation of a CD3/CD19 depleted stem cell grafts after dose reduced conditioning for the treatment of treatment refractory or relapsed hematologic malignancies after preceding allogeneic or autologous hematopoietic cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age <60, >18 years
* Karnofsky >60%
* High risk hematologic malignancy or relapse after preceding auto/allo HCT in patients with:
* ALL
* AML
* PNH
* MDS (RAEB-t/secondary AML)
* NHL
* ALL
* HD
* CML
* MM
* No HLA-identical MRD or URD if not preceding allo-HCT
* Use haploidentical donor with KIR-Mismatch if choice

Exclusion Criteria:

* < 3 months after preceding HCT
* Active cerebral seizures
* > 30% blasts in BM if ALL/AML/CML-BC
* Completely chemo-refractory
* Preceding myocardial infarction
* Ejection fraction <30 % echocardiography
* Creatinine clearance <50 ml/min
* Respiratory insufficiency on supplemental O2 or DLCO < 30%
* Allergy against murine antibodies
* HIV infection
* Pregnancy
* Unable for informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2004-02; Primary Completion 2009-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Engraftment
Toxicity
Mortality and Morbidity

SECONDARY OUTCOMES:
Infections
GVHD
Immune reconstitution
Disease response
Long term toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang A Bethge, MD, Principal Investigator — University of Tuebingen Medical Center
Locations (7):
- Germany (7):
  - University of Dresden Medical Center, Dresden
  - Center for Marrow Transplantation, Essen
  - Medical Center University of Hamburg, Hamburg
  - Medical Center University of Muenster, Münster
  - South West German Cancer Center, University of Tuebingen Medical Center, Tübingen
  - Deutsche Klinik für Diagnostik, Wiesbaden
  - University of Wuerzburg Medical Center, Würzburg

REFERENCES:
- [Derived] Federmann B, Bornhauser M, Meisner C, Kordelas L, Beelen DW, Stuhler G, Stelljes M, Schwerdtfeger R, Christopeit M, Behre G, Faul C, Vogel W, Schumm M, Handgretinger R, Kanz L, Bethge WA. Haploidentical allogeneic hematopoietic cell transplantation in adults using CD3/CD19 depletion and reduced intensity conditioning: a phase II study. Haematologica. 2012 Oct;97(10):1523-31. doi: 10.3324/haematol.2011.059378. Epub 2012 Apr 4. PMID 22491731
- See also: Related Info — http://www.onkologie-tuebingen.de